CLINICAL TRIAL: NCT06660979
Title: Using Reinforcement Learning to Personalize Electronic Health Record Tools to Facilitate Deprescribing
Acronym: REINFORCE-EHR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Atrius Health (Other)
Responsible Party: Principal Investigator, Julie Lauffenburger, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2024P002700; 2P30AG064199-06 (NIH)
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Aging
Keywords: Medication optimization; High-risk medications
MeSH Terms: interventions — Reinforcement Machine Learning

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reinforcement learning intervention (Experimental): The intervention is a reinforcement learning program that personalizes EHR-based tools for PCPs to promote deprescribing high-risk medications over follow-up. The reinforcement learning intervention selects a tool for each provider based on an algorithm from an inventory of EHR tools and chooses tools that are predicted to motivate action for the individual provider. The effectiveness of each tool will be assessed on a selected interval based on whether a deprescribing action is taken by PCPs for eligible patients. The algorithm is trained to maximize these actions over time.
  Interventions: Behavioral: Reinforcement learning
- Usual care (No Intervention): No EHR-based tools provided beyond those used in regular clinical practice.

INTERVENTIONS:
Behavioral: Reinforcement learning — The intervention is a reinforcement learning program that personalizes EHR-based tools for PCPs to promote deprescribing high-risk medications over follow-up. The reinforcement learning intervention selects a tool for each provider based on an algorithm from an inventory of EHR tools and chooses tools that are predicted to motivate action for the individual provider. The inventory of EHR tools from which the algorithm will choose include the following potential factors: open encounter, order entry, cold-state outreach, simplification, and risk framing.
  Arms: Reinforcement learning intervention

SUMMARY:
The overall goal of the proposed research is to refine and adapt and perform efficacy testing of a novel reinforcement learning-based approach to personalizing EHR-based tools for PCPs on deprescribing of high-risk medications for older adults. The trial will be conducted at Atrius Health, an integrated delivery network in Massachusetts, and will intervene upon primary care providers. The investigators will conduct a cluster randomized trial using reinforcement learning to adapt electronic health record (EHR) tools for deprescribing high-risk medications versus usual care. 70 PCPs will be randomized (i.e., 35 each to the reinforcement learning intervention and usual care [no EHR tool] in each arm) to the trial and follow them for approximately 30 weeks. The primary outcome will be discontinuation or ordering a dose taper for the high-risk medications for eligible patients by included primary care providers, using EHR data at Atrius. The primary hypothesis is that the personalized intervention using reinforcement learning will improve deprescribing compared with usual care.

ELIGIBILITY:
Inclusion Criteria:

The trial will intervene upon primary care providers (including physicians and PCP-designated nurse practitioners and physician assistants) at Atrius Health.

Patients of the PCPs will be included in the intervention and analysis if they are >/=65 years of age and have been prescribed >/= 90 pills of high-risk medications in the prior 180 days based on EHR data.

Exclusion Criteria:

• Not a primary care provider at Atrius Health

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Discontinuation or taper for high-risk medication | Through trial completion, up to 7 months
  Deprescribing will be assessed using routinely collected data from the EHR system for eligible patients flagged as in need of deprescribing. The deprescribing outcome will be a "reduction" in inappropriate prescribing, defined as either discontinuation of one the the medication classes of interest or ordering a dose taper.

SECONDARY OUTCOMES:
Discontinuation of high-risk medication | Through trial completion, up to 7 months
  Discontinuation of medication assessed using routinely-collected data from the EHR system for eligible patients flagged as in need of deprescribing.

CONTACTS AND LOCATIONS:
Locations (1):
- Atrius Health, Boston, Massachusetts, United States